CLINICAL TRIAL: NCT06340295
Title: A Multicenter, Prospective Cohort Study of Preserved Ratio Impaired Spirometry(PRISm) in a Population
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Shanxi Bethune Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Tianjin Medical University General Hospital (Other); The First Hospital of Qinhuangdao (Other Government); Shandong Provincial Hospital (Other Government); Second Hospital of Jilin University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); MinDong Hospital of Ningde City (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023313
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: COPD
Keywords: PRISm; COPD; Imaging omics; Metabolomics; proteomics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- new-onset COPD group: FEV1/FVC<0.7 after bronchodilator inhalation during 3 years of follow-up
- Continuous PRISm group: After bronchodilator inhalation, FEV1/FVC≥70% and the percentage of FEV1pred%<80% during 3 years of follow-up
- PRISm to normal group: After bronchodilator inhalation, FEV1/FVC≥0.7 and FEV1pred% ≥80% during 3 years of follow-up

INTERVENTIONS:
Other:

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the most common chronic tract disease and the third leading cause of death worldwide. The treatment effect of COPD is poor, and the disease is progressive, resulting in a serious disease burden. The key reason is that early recognition is difficult and the early pathophysiological mechanism is unclear, which leads to the difficulty of early intervention.PRISm is likely to be the precursor stage of COPD, which may provide an important research object for the study of pathophysiological characteristics, inflammation and immunomodulatory mechanisms of early COPD, and may also become a new entry point for early intervention of COPD. This study attempts to establish a PRISm prospective cohort，and collects blood, EBC and urine for analysis of inflammatory factors, metabolomics, proteomics and microbiome, and performs chest HRCT to obtain imaging indicators, and conducts 3-year dynamic follow-up observation to study the evolution characteristics of pulmonary function and the incidence of COPD in the PRISm cohort. To compare the differences in imaging, inflammatory factors, metabolomics, proteomics and microbiome among the three PRISm groups, and establish a risk prediction model for progression to COPD through PRISm. It lays a foundation for understanding the characteristics of COPD at an earlier stage and exploring new early warning indicators.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age range from 20 to 75 years old, regardless of gender; 2) Pulmonary function test: After inhaling bronchodilators, FEV1/FVC ≥ 70%, and FEV1<80% of the expected value; 3) Agree to enter this research project and sign an informed consent form 4) Able to comply with research protocols.

Exclusion Criteria:

* 1) Confirmed chronic obstructive pulmonary disease, bronchial asthma, bronchiectasis, interstitial lung disease, occupational lung disease, tuberculosis, pulmonary vascular disease, central airway stenosis and other confirmed respiratory diseases.

  2) Have undergone lobectomy and/or lung transplantation; 3) complicated with serious underlying diseases (including serious mental illness, mental retardation, neurological disease, malignant tumor, chronic liver disease, heart failure, autoimmune disease, chronic kidney disease); 4) accompanied by severe pleural disease and/or lesions of the sternum or ribs; 5) Have active tuberculosis or are receiving anti-tuberculosis treatment; 6) Pregnancy or lactation; 7) Can not be followed up for a long time or poor compliance;

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects are 1430 PRISm people from the PIFCOPD cohort in our center and 600 newly enrolled PRISm people in this study, totaling approximately 2000 PRISm people.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The number and proportion of newly diagnosed COPD | the third year of follow-up
  FEV1/FVC<0.7 after bronchodilator inhalation during 3 years of follow-up

SECONDARY OUTCOMES:
The number and proportion of continuous PRISm population | the third year of follow-up
  After bronchodilator inhalation, FEV1/FVC≥70% and the percentage of FEV1pred%<80% during 3 years of follow-up
The number and proportion of PRISm to normal population | the third year of follow-up
  After bronchodilator inhalation, FEV1/FVC≥0.7 and FEV1pred% ≥80% during 3 years of follow-up
Emerging diseases | the third year of follow-up
  Emerging diseases: non-COPD lung diseases (bronchial asthma, ILD), OSA, cardiovascular diseases (such as coronary heart disease, hypertension, etc.), endocrine diseases (such as diabetes), cerebrovascular diseases, digestive diseases, chronic kidney diseases, etc.
Death and cause of death | the third year of follow-up
  Death and cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD., Study Chair — Peking University First Hospital
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Shandong Provincial Hospital Affiliated to Shandong University, Jing’an
  - Shanxi Bethune Hospital, Taiyuan

IPD SHARING:
Plan to Share IPD: No